CLINICAL TRIAL: NCT03458000
Title: Capsule Endoscopy for Hemorrhage in the ER
Acronym: CHEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Andrew Meltzer, Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ISR-2016-10770; IRB #041707 (Other: George Washington University Institutional Review Board); NCT01371591 (obsolete NCT alias)
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: capsule endoscopy; PillCam; upper Endoscopy; emergency Department; upper gastrointestinal bleeding; GI bleed
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Control (Active Comparator): Video Capsule Endoscopy will be administered during ED, but video will not be read until after inpatient EGD. Subject will have hospital admission with an EGD conducted during hospital stay.
  Interventions: Other: Standard of Care
- Experimental (Experimental): Subject will have Video Capsule Endoscopy read during ED length of stay, disposition will be determined using Capsule Endoscopy Risk Assessment.
  Interventions: Device: PillCam UGI

INTERVENTIONS:
Device: PillCam UGI — An esophageal capsule endoscope which is designed to visualize the upper gastrointestinal tract.
  Arms: Experimental
Other: Standard of Care — Patient was admitted to hospital for care and received in-patient EGD.
  Other Names: SOC
  Arms: Active Control

SUMMARY:
This is a multi-center randomized controlled trial examining the use of Video Capsule Endoscopy (VCE) to discharge low-moderate risk patients with suspected upper gastrointestinal bleeds (UGIB) from the Emergency Department (ED.) The investigators will enroll 100 subjects at 4 sites who present with signs of hemodynamically stable UGIBs and compare VCE risk assessment to an Active Control (AC) group who receive inpatient upper endoscopy (EGD).

DETAILED DESCRIPTION:
Video capsule endoscopy (VCE) was initially approved in 2001 by the Food and Drug Administration. VCE offers potential advantages over traditional EGD including the ability to be performed 24 hours a day without sedation and interpreted at the bedside by emergency physicians. In addition, VCE is much less invasive, is painless, and enables the patient to pursue normal daily activities after the procedure.

Our primary goal is to test whether ED Video Capsule Endoscopy (VCE) is able to safely discharge low risk patients for outpatient evaluation and management. Our secondary objective is to estimate the sensitivity and specificity of VCE compared to subsequent EGD in the detection of serious bleeding lesions in the upper gastrointestinal (GI) tract.

Research Coordinator will screen potential patients with signs of upper GI bleeding. Patients who screen as eligible will be approached about potential interest, to review of inclusion and exclusion criteria, and obtain informed consent. Research Coordinator will calculate traditional risk stratification scores and once enrolled, all subjects will be randomized to either Active Control (AC) [admission plus EGD within hospital stay] or experimental Capsule Endoscopy Risk Assessment (CERA) in ED. Only patients randomized to the experimental arm will receive video capsule endoscopy in the emergency department.Within 2 hours of presenting to the ED, patient will ingest video capsule-- RC will monitor progress on real-time viewer for passage through pylorus. Upon passing the pylorus, we will record 5 more minutes of video or until battery runs out - whichever occurs first. Patient data will be completed using a standardized data collection tool including the following elements: chief complaint of patient, history of present illness, past medical history, pertinent lab findings, current medications, vital signs, focused physical exam findings and all relevant treatments administered during the ED and hospital stay.

For Active Control (AC) group each patient will be admitted. During hospital admission, EGD will be performed on all subjects and hemostasis therapy applied as necessary. The study team decided against mandating that EGD be performed within 24 hours of hospital admission.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged ≥ 18 years presenting to the Emergency Department with likely upper GI bleed (bloody emesis and/or coffee ground vomiting and/or melena) that has occurred within the previous 48 hours.

Exclusion Criteria:

1. Upper GI Bleed with hemodynamic instability (BP<90 mmHg, pulse>120 beats per minute, and Hgb < 9 g/dL)
2. High Risk Upper GI Bleed (Glasgow Blatchford Score* ≥ 6)
3. Signs, symptoms or history of liver cirrhosis or liver failure
4. Signs, symptoms or history of decompensated heart failure or congestive heart failure
5. Presumed Pregnant, trying to conceive or breastfeeding
6. Known history of gastric cancer
7. Known history of gastric or esophageal varices
8. GI surgery within the last 6 months
9. Prior enrollment in the CHEER Study
10. Prisoner or Ward of State
11. Trouble swallowing, suspected bowel obstruction or perforation, per treating clinician
12. Past UGI tract surgery (e.g., Bilroth I or II, esophagectomy, gastrectomy, bariatric procedure) that changes Gastrointestinal anatomy
13. Known history of gastroparesis, esophageal stricture or Crohn's disease
14. Altered mental status that limits the ability to swallow a capsule
15. Expected to have Magnetic Resonance Imaging (MRI) examination within 7 days
16. Consumed medications within the past 12 hours that may coat the upper GI tract such as antacids or sucralfate or Maalox and potentially limits capsule visualization
17. Patient either refuses or is unable to get traditional EGD
18. Patient does not have reliable contact information - no phone, no permanent address
19. Patient refuses
20. Unable to provide written consent
21. Non-English speaker
22. Suspected middle or lower GI bleeding
23. Treating ED Physician is not amenable to admission or discharge based on randomization or Video Capsule Endoscopy results. * As a modification, the GBS Score modified from the traditional GBS score to reduce the Hemoglobin cut-off for 6 points from 10g/dL to 9 g/dL (see Appendix B, CHEER 4; patient screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Meltzer, MD, Principal Investigator — George Washington University- Department of Emergency Medicine
Locations (3):
- United States (3):
  - George Washington University, Washington D.C., District of Columbia
  - Duke University School of Medicine, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meltzer AC, Ali MA, Kresiberg RB, Patel G, Smith JP, Pines JM, Fleischer DE. Video capsule endoscopy in the emergency department: a prospective study of acute upper gastrointestinal hemorrhage. Ann Emerg Med. 2013 Apr;61(4):438-443.e1. doi: 10.1016/j.annemergmed.2012.11.008. PMID 23398660

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Control | Experimental
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Control | Experimental | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47.0 [41.0 to 54.0] | 55.0 [36.0 to 58.0] | 51.5 [38.5 to 57.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 7 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 7 | 9 | 16
  Race: Other | 2 | 0 | 2
  Race: White | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Discharged for Outpatient Management of Upper GI Bleeds
Description: Our primary goal is to determine whether ED VCE is able to discharge low risk patients for outpatient management of upper GI bleeds.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Active Control | Experimental
Number analyzed (Participants) | 13 | 11
Participants | 3 | 9

2. Secondary Outcome: Detection Rate of Video Capsule Endoscopy
Description: Our secondary objective is to present the prevalence of clinical findings in VCE subjects based on gastroenterologist interpretation.
Time Frame: 30 Days
Population: This is a subgroup analysis. The reason only the experimental arm is reported here is because only the experimental arm got the VCE.
Measure: Number; unit: participants
Groups:
- Experimental: Video Capsule Endoscopy (VCE) Arm
Arm/Group | Experimental
Number analyzed (Participants) | 11
participants
  Clean stomach and duodenum i.e. no fresh blood /coffee grounds | 8
  Upper GI pathology non-causative/ incidental. | 1
  A low grade non-Variceal lesion (Forrest IIc, III) | 1
  Coffee ground blood | 2
  Fresh blood or evidence of active bleeding | 1
  Other sources of non-variceal bleeding / pathology | 3
  VCE passed the pylorus | 9
  Needs endoscopic hemostasis | 2

3. Other Pre Specified Outcome: Patient Satisfaction With VCE Procedure
Time Frame: 30 Days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: GI Physician Final Read and Site Physician Agreement on VCE Results
Time Frame: 30 Days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events at Day 7 and Day 30
Description: Assess for mortality, re-bleeding, total blood transfusions, surgery (capsule-specific group)
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Active Control | Experimental
Number analyzed (Participants) | 13 | 11
Participants | 0 | 0

6. Other Pre Specified Outcome: ED Length of Stay
Time Frame: 30 Days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Hospital Length of Stay
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious Adverse Events, and Other Adverse Events were monitored/assessed at Day 7 and Day 30
Description: No adverse events were elicited at day 7 or day 30
Arm/Group | Active Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT03458000/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03458000/ICF_001.pdf